CLINICAL TRIAL: NCT04973787
Title: MicroSpA & MicroRA: The Role of Microbiome on Biological Therapy Efficacy in Axial Spondyloarthritis and Rheumatoid Arthritis - a New Paradigm
Brief Title: The Role of Microbiome on Biological Therapy Efficacy in axSpA and RA
Acronym: MicroSpA & RA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Centro Hospitalar Lisboa Ocidental Hospital Egas Moniz (Unknown); Centro Hospitalar De São João, E.P.E. (Other); Centro Hospitalar de Vila Nova de Gaia/Espinho (Other); Centro Hospitalar Universitário de Lisboa Norte - Hospital de Santa Maria (Unknown); Instituto Português de Reumatologia (Unknown); Centro Hospitalar Médio Tejo - Hospital Rainha Santa Isabel - Torres Novas (Unknown); Centro Hospitalar Baixo Vouga - Hospital Infante D. Pedro (Unknown); Comprehensive Health Research Center (Other); iNOVA4Health - Rheumatic Diseases Lab (Unknown); Unidade Local de Saúde do Alto Minho, Hospital Conde de Bertiandos (Unknown); Hospital de Braga E.P.E. (Unknown); Hospital Sousa Martins - Unidade de Saúde Local da Guarda (Unknown)
Responsible Party: Sponsor
Other Study IDs: MicroSpA
Record Dates: First submitted 2021-06-22; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Axial Spondyloarthritis; Arthritis, Rheumatoid
Keywords: Tumor Necrosis Factor alpha inhibitor; Microbiota; Biomarker
MeSH Terms: conditions — Axial Spondyloarthritis; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- axSpA: Patients with clinical diagnosis of axialSpondyloarthritis according to ASAS criteria, with indication for bDMARD (Portuguese Rheumatology Society Guidelines)
  Interventions: Biological: biological disease-modifying antirheumatic drugs (bDMARDs)
- RA: Patients with clinical diagnosis of Rheumatoid arthritis according to 2010 ACR/EULAR classification criteria, with indication for bDMARD (Portuguese Rheumatology Society Guidelines)
  Interventions: Biological: biological disease-modifying antirheumatic drugs (bDMARDs)
- Control: Healthy participants, e.g. with no clinical diagnosis of rheumatic inflammatory disease, crossed by age, gender and diet profile

INTERVENTIONS:
Biological: biological disease-modifying antirheumatic drugs (bDMARDs) — bDMARD therapy (TNF inhibitors), according to the Portuguese recommendations for the use of biological therapies in patients with axSpA and RA
  Groups: RA; axSpA

SUMMARY:
Spondyloarthritis (SpA) and Rheumatoid arthritis (RA) are among the most common chronic inflammatory rheumatic diseases. Introduction of Tumor Necrosis Factor alpha inhibitors (TNFi) to the therapeutic strategy improved acute inflammation and pain, but a significant percentage of patients develop severe adverse events or are still non responders or incomplete responders to these expensive treatments. There is an urgent need to identify new predictors of biological therapy response. It has been described the role of microbiota in some rheumatic diseases, however, clinical trials are scarce. We hypothesized that microbiota or their metabolites may play a role in therapeutic response to TNFi.

DETAILED DESCRIPTION:
Thus, this project aimed to evaluate the influence of oral and gut microbiota in the therapeutic response to biologic therapies, in 60 patients.

It is expected to enrolled 30 SpA and 30 RA patients and 30 controls, crossed by gender, age and diet profile. Oral and fecal microbiota will be characterized before TNFi therapeutic. Patients will have an additional microbiota and metabolic profile characterization 14 weeks late after.

This will allow to identify specific profiles of oral and gut microbiome and/or specific biochemical patterns in these patients. At week 14 it will be possible to identify changes induced by TNFi. In addition, it will be possible to identify microbiota pattern associated clinical therapeutic TNFi response vs non-response.

This will allow to predict isolate microbe or microbes patterns at baseline associated to clinical response obtained at week 14. These results may additionally contribute to clinical decision and a better evidenced-based treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of axSpA (according to ASAS classification criteria) or RA (according to 2010 ACR/EULAR classification criteria);
2. Indication for bDMARD therapy, according to the Portuguese recommendations for the use of biological therapies in patients with axSpA and RA;
3. Oral corticosteroids (equivalent to prednisolone ≤ 10mg/day) and/or nonsteroidal anti-inflammatory drugs allowed at stable dose ≥4 weeks before baseline;
4. Conventional DMARDs allowed at stable dose ≥12 weeks before baseline;
5. Ability to provide informed consent.

Exclusion Criteria:

1. History of rheumatic disorder other than axSpA or RA;
2. History of Inflammatory Bowel Disease;
3. Previous treatment with bDMARD;
4. Current pregnancy or breastfeeding;
5. Malignancy (except for completely treated squamous or basal cell carcinoma);
6. Any uncontrolled medical condition (e.g., uncontrolled diabetes mellitus, unstable ischemic heart disease);
7. History of any documented gastrointestinal disease or tract surgery leaving permanent residua (e.g., gastrectomy, bariatric surgery, or colectomy);
8. Intraarticular injections of extra-axial joints and tendons within 28 days before or at baseline;
9. Recent (<3 months prior) use of any antibiotic therapy, current extreme diet (e.g., parenteral nutrition or macrobiotic diet), current consumption of probiotics.

Control group will be healthy participants, and the same inclusion and exclusion criteria will be applied except for rheumatic disease diagnosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with axSpA or RA according to ASAS and 2010 ACR/EULAR classification criteria, respectively, with indication to start bDMARD according to Portuguese Rheumatology Society.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Oral and gut microbiota characterization in axSpA and RA patients at baseline | Before bDMARD
Oral and gut microbiota characterization in axSpA and RA patients at week 14 | 14 weeks after start bDMARD
Disease activity measured by ASAS20 in axSpA and ACR20 in RA | 14 weeks after start bDMARD

SECONDARY OUTCOMES:
Changes in Erythrocyte Sedimentation Rate (ESR, measured in mm/h) | Before bDMARD and 14-week after start bDMARD
Changes in High-sensitivity C-reactive protein (hsCRP, measured in mg/dL) | Before bDMARD and 14-week after start bDMARD
Disease activity characterization using Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) in axSpA | Before bDMARD and 14-week after start bDMARD
  Scale from 0 (worse outcome) to 10 (better outcome)
Disease activity characterization using Ankylosing Spondylitis Disease Activity Score - C-Reactive Protein (ASDAS-CRP) in axSpA | Before bDMARD and 14-week after start bDMARD
  < 1.3 Inactive disease; > 3.5 Very high disease activity
Disease activity characterization using Disease Activity Score-28 for Rheumatoid Arthritis with C-Reactive Protein (DAS28-CRP) for RA | Before bDMARD and 14-week after start bDMARD
  Score greater than 5.1 implies active disease, less than 3.2 low disease activity, and less than 2.6 remission
Quality of life evaluation with Short form 36 (SF36) at baseline and week 14 | Before bDMARD and 14-week after start bDMARD
  Score from 0 (worse outcome) to 100 (better outcome)
Quality of life evaluation with Ankylosing Spondylitis Quality of Life (ASQOL) at baseline and week 14 | Before bDMARD and 14-week after start bDMARD
  Range from 0 -18 - High scores indicate worse quality of life
Quality of life evaluation with Health Assessment Questionnaire (HAQ) at baseline and week 14 | Before bDMARD and 14-week after start bDMARD
  Scores of 0 to 1 are generally considered to represent mild to moderate difficulty, 1 to 2 moderate to severe disability, and 2 to 3 severe to very severe disability
Quality of life evaluation regarding depression and anxiety using Hospital Anxiety and Depression Scale (HADS) at baseline and week 14 | Before bDMARD and 14-week after start bDMARD
  Scores of less than 7 indicate non-cases; 8-10 Mild; 11-14 Moderate;15-21 Severe
Fatigue evaluation at baseline and week 14 | Before bDMARD and 14-week after start bDMARD
  Visual analogic scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Faria, PhD, Principal Investigator — Universidade Nova de Lisboa; Fernando Pimentel-Santos, PhD Agg, Principal Investigator — NOVA Medical School, Universidade NOVA de Lisboa; CHLO Hospital Egas Moniz
Locations (10):
- Portugal (10):
  - Centro Hospitalar Baixo Vouga - Hospital Infante D. Pedro, Aveiro
  - Hospital de Braga, E.P.E., Braga
  - Hospital Sousa Martins - Unidade de Saúde Local da Guarda, Guarda
  - Centro Hospitalar Lisboa Ocidental - Hospital Egas Moniz, Lisbon
  - Centro Hospitalar Universitário de Lisboa Norte - Hospital Santa Maria, Lisbon
  - Instituto Português de Reumatologia, Lisbon
  - Unidade Local de Saúde do Alto Minho, Hospital Conde de Bertiandos, Ponte de Lima
  - Centro Hospitalar Universitário São João, Porto
  - Centro Hospitalar de Médio Tejo - Hospital Rainha Santa Isabel - Torres Novas, Torres Novas
  - Centro Hospitalar de Vila Nova da Gaia/Espinho, Vila Nova de Gaia

IPD SHARING:
Plan to Share IPD: No